CLINICAL TRIAL: NCT01414231
Title: Randomised Comparison of OSHO Induction vs. the German AML Intergroup Standard, Randomised Comparison of AraC/Mtx vs. Flu/AraC/Mtx in Pts Without CR After One Induction Cycle and Randomized Comparison of One vs. Two Consolidation Therapies.
Brief Title: Comparison of the OSHO Protocol to a Standard Arm Protocol of the German AML Intergroup in Patients With AML<60a
Acronym: OSHO#061
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Prof. Dr. med. Dr. h. c. Dietger Niederwieser, University of Leipzig, Hematology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML 2002 #061
Record Dates: First submitted 2011-08-05; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2008-04

CONDITIONS: Acute Myeloid Leukaemia
Keywords: AML; acute myeloid leukaemia; low vs intermediate dose AraC; CR rate; patients <60 years
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cytarabine low dose (Active Comparator): This is the golden standard of AML treatment
  Interventions: Drug: Cytarabine
- Cytarabine intermediate dose (Active Comparator): This is the OSHO internal arm
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — Intermediate dose against low dose; IDA 12 mg/m2 iv days 1 - 3 and AraC 2 x 1 g/m2 bid on days 1+3+5+7 vs. AraC 100 mg/m2/day i.v.-for 7 days and Daunorubicin 60 mg/m2/Tag on days 3, 4 und 5.

SUMMARY:
This protocol is part of the German AML Intergroup Trial, where the OSHO study arm is compared to the common German standard arm after randomization in a 9:1 ratio. The hypothesis involves primarily dosing and application of AraC for induction. It is expected that CR rates and as a consequence also LFS are higher in protocols using higher AraC compared to lower doses and that LFS might be superior in the study specific arm compared to the golden standard published several years ago. In the standard arm, AraC 100mg/m2/day is given as continuous infusion over 7 days. Daunorubicin is given as 60 mg/m2/day over a two hours infusion on days 3, 4 und 5. On day 22 a second induction course is applied. After reaching CR, three cycles of AraC 3 g/m2 over three hours bid are infused on day 1, 3 und 5. In contrast the OSHO arm consists of induction therapy with IDA 12 mg/m*2 over 20-30-min-iv on day 1 - 3 and AraC 2 x 1 g/m*2 bid over 3-h-iv on days 1+3+5+7.

A previous phase II study of the OSHO has shown high CR in patients with relapsed AML using MitoFlag. In this study we asked the question if MitoFlag is superior to IdaAraC in newly diagnosed AML patients without CR after the first induction chemotherapy. Therefore patients are randomized to receive either MitoFlag or IdaAraC and the difference in CR rates evaluated.

It is still unclear if two consolidation therapies are needed before allogeneic or autologous stem cell transplantation. This question is being addressed in the second part of the OSHO study, where patients are randomized to receive either one or two consolidation therapies.

In this study all patients with AML and an age of 18-60 years except M3 are entered

ELIGIBILITY:
Inclusion Criteria:

Adult patients < or = 60 years acute myelogenous leukemia (AML) AML t(8;21)(q22;q22), AML1 (CBFa)/ETO, AML(inv(16)(p13q22)) und variants (CBFb/MYH11), AML 11q23, MLL-anomalies, AML with normal karyotyp myelodysplastic syndrome (MDS)RAEBT with 20-30% blasts.

de novo AML secundary AML after MDS secundary AML after chemotherapy with alkylantien sekundäre AML after chemotherapy with Epipodophyllotoxin informed consent

Exclusion Criteria:

AML M3 patients included in another clinical trial contraindications for high dose cytotoxic therapy such as renal insufficiency liver insufficiency cardiac insufficiency NYHA III + IV, acute myocardial infarction uncontroled infection like pneumonia with hypoxemia or septic schock pregnancy Karnofski-Index of 10 and less second maligancy severe, decompensated metabolism disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 850 (Estimated)
Dates: Start 2002-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Event free survival | after 5 years

SECONDARY OUTCOMES:
Complete remission | average of 6 weeks
Overall survival | at 5 years average
Relapse free survival | at 5 years average

CONTACTS AND LOCATIONS:
Overall Officials: Dietger Niederwieser, MD, Principal Investigator — University of Leipzig
Locations (1):
- University of Leipzig, Hematology, Leipzig, Germany

REFERENCES:
- [Derived] Buchner T, Schlenk RF, Schaich M, Dohner K, Krahl R, Krauter J, Heil G, Krug U, Sauerland MC, Heinecke A, Spath D, Kramer M, Scholl S, Berdel WE, Hiddemann W, Hoelzer D, Hehlmann R, Hasford J, Hoffmann VS, Dohner H, Ehninger G, Ganser A, Niederwieser DW, Pfirrmann M. Acute Myeloid Leukemia (AML): different treatment strategies versus a common standard arm--combined prospective analysis by the German AML Intergroup. J Clin Oncol. 2012 Oct 10;30(29):3604-10. doi: 10.1200/JCO.2012.42.2907. Epub 2012 Sep 10. PMID 22965967